CLINICAL TRIAL: NCT06655350
Title: Is Harvesting the Peroneus Brevis an Alternative in Anatomic Ankle Ligament Reconstruction
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: IRBN752024/CHUSTE
Record Dates: First submitted 2024-10-22; First posted 2024-10-23 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Ankle Disease; Ankle (Ligaments); Instability (Old Injury)
Keywords: Ankle instability; Graft; Peroneus brevis; Ankle ligament reconstruction
MeSH Terms: interventions — Weights and Measures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Harvested ankle
  Interventions: Other: MRI; Other: Measure
- Native ankle
  Interventions: Other: MRI; Other: Measure

INTERVENTIONS:
Other: MRI — Morphological data on the tendon (appearance) will be collected on the harvested side and on the healthy side from an MRI analysis carried out systematically after Haemi-Castaing-type surgery.
Other: Measure — Morphological data on the tendon (diameter) will be collected on the harvested side and on the healthy side from an MRI analysis carried out systematically after Haemi-Castaing-type surgery.

SUMMARY:
Severe ankle sprains are the most frequent reason for emergency trauma consultations. Between 30% and 80% of sprains result in sequelae such as pain, joint derangement or instability. Ankle instability can itself lead to osteoarthritis if left untreated (1st cause of post-traumatic ankle osteoarthritis). To treat instability, ligament reconstruction is performed by harvesting the tendon of the gracilis muscle (inserted at knee level) to replace the damaged ankle ligaments. This tendon is also used for other ligament reconstructions (anterior cruciate ligament), so is not always harvested. Moreover, it represents an invasive procedure at a distance from the site of interest (the ankle), and can cause sensory nerve damage (20-60% of cases). For a long time, half of the peroneus brevis tendon was harvested as part of a now-defunct ankle stabilization technique (Hemi-Castaing). This tendon does, however, play a role in stabilizing the ankle.

DETAILED DESCRIPTION:
Before considering harvesting the peroneus brevis as an alternative to harvesting the gracilis, it is important to ensure that the peroneus brevis remains functional after harvesting. The aim of this study was to evaluate the potential for tendon regrowth after harvesting half of the peroneus brevis tendon after Hemi-Castaing-type ankle stabilization surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult one year after peroneus brevis harvesting (Hemi-Castaing)

Exclusion Criteria:

* No.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at Saint-Etienne University Hospital who underwent Haemi-Castaing-type ankle stabilisation surgery.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2024-09-06 (Actual); Primary Completion 2024-10-11 (Actual); Study Completion 2024-10-11 (Actual)

PRIMARY OUTCOMES:
Peroneus brevis diameter of a native ankle and at one-year postoperative harvested ankle. | Year : 1
  Cross section area (mm²) at 40, 30, 20mm above the tip of the fibula, and 20mm from 5th metatarsal basis.

SECONDARY OUTCOMES:
Peroneus brevis MRI aspect of a native ankle and at one-year postoperative harvested ankle. | Year : 1
  % T1 signal on the tendon at 40, 30, 20mm above the tip of the fibula, and 20mm from 5th metatarsal basis.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Henri Vermorel, MD, Principal Investigator — CHU de Saint-Etienne
Locations (1):
- CHU de Saint-Etienne, Saint-Priest-en-Jarez, France

IPD SHARING:
Plan to Share IPD: No